CLINICAL TRIAL: NCT06232369
Title: Research on Threat Reversal Abnormality and Underlying Neural Mechanisms in Patients With Anxiety Disorders
Brief Title: Threat Reversal Abnormality in Patients With Anxiety Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Kangning Hospital (Other)
Collaborators: The National Natural Science Foundation of China (NSFC) (Unknown)
Responsible Party: Principal Investigator, Jingchu Hu, Associate Research Fellow, Shenzhen Kangning Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 82201672
Record Dates: First submitted 2024-01-10; First posted 2024-01-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Anxiety Disorder; Anxiety State
Keywords: Threat Reversal; Emotion Flexibility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient group + active stimulation intervention (Experimental): Patient participants with anxiety disorders in this arm will first accept active repetitive stimulation on core brain regions and then complete the threat reversal learning paradigm.
  Interventions: Device: Active repetitive deep transcranial magnetic stimulation (dTMS)
- Patient group + sham stimulation intervention (Sham Comparator): Patient participants with anxiety disorders in this arm will first accept sham repetitive stimulation on core brain regions and then complete the threat reversal learning paradigm.
  Interventions: Device: Sham repetitive deep transcranial magnetic stimulation (dTMS)
- Healthy control group + sham stimulation intervention (Sham Comparator): Healthy participants in this arm will first accept sham repetitive stimulation on core brain regions and then complete the threat reversal learning paradigm.
  Interventions: Device: Sham repetitive deep transcranial magnetic stimulation (dTMS)

INTERVENTIONS:
Device: Active repetitive deep transcranial magnetic stimulation (dTMS) — Before the intervention, the brain structure of each participant will be captured using an MRI scanner, and individualized spatial coordinates of the hypothesized target will be determined based on these 3D structural images. Then the resting motor threshold will be tested using the method of thumb twitching observation.
  The intervention will employ the H7 coil that is accurately delivered to the intended target by an optic navigation and a deep pulse protocol at 90% of the tested threshold for 15-minute stimulation duration.
  Arms: Patient group + active stimulation intervention
Device: Sham repetitive deep transcranial magnetic stimulation (dTMS) — Before the intervention, the brain structure of each participant will be captured using an MRI scanner, and individualized spatial coordinates of the hypothesized target will be determined based on these 3D structural images. Then the resting motor threshold will be tested using the method of thumb twitching observation.
  The intervention will employ the H7 coil that is placed on the scalp to mimic the sensation and sounds of the actual treatment but without letting the magnetic field reach the brain tissue for 15-minute duration.
  Arms: Healthy control group + sham stimulation intervention; Patient group + sham stimulation intervention

SUMMARY:
The goal of this clinical trial is to explore the flexibility of threat control and underlying neural mechanism based on the threat reversal paradigm (a highly validated new paradigm where threat learning and inhibition are required) in patients with anxiety disorders (mainly generalized anxiety disorder). The hypotheses are:

1. Threat reversal abilities are hypothesized to be impaired in patients with anxiety disorders compared to healthy normal subjects, which are assumed to be associated with anxiety symptoms.
2. The neural mechanism underlying threat reversal abnormalities in patients with anxiety disorders is hypothesized to involve the prefrontal cortex, amygdala, and hippocampus.
3. The repetitive stimulation to the core brain regions of threat reversal is assumed to improve threat reversal abilities and anxiety symptoms of patients.

DETAILED DESCRIPTION:
In this study, there are three sub-trials in combination with skin conductance response (SCR), functional magnetic resonance imaging (fMRI), and non-invasive neuromodulation techniques to uncover the abnormal threat reversal in anxiety disorder at behavioral and neural levels.

Participants in the first trial will learn the threat of emotional faces based on the Pavlovian conditioned fear learning paradigm; their neural activities in the hypothesized brain regions will be obtained via brain imaging equipment. The researchers will compare the differences among three groups (one patient group, two healthy control groups with different anxiety level) on performance in the threat reversal task, and their neural activities and brain functional connectivity characteristics, in order to reveal the potential behavioral threat reversal abnormalities and core associated brain regions underlying threat reversal.

Participants in the second trial will be given the same learning paradigm and brain imaging equipment as in the first, but with repetitive stimulation intervention on the core brain regions determined in study 1. Using a double-blind randomized controlled experiment, the participants will be divided into three groups (active stimulation + patient, sham stimulation + patient, and sham stimulation + healthy control). The researchers will compare the behavioral differences in the threat reversal task after active and sham stimulation.

Participants in the third trial will be given the same study design and intervention as the second trial, but for eight weeks. Finally, the researchers will retest and compare the improvement in threat reversal abilities and anxiety symptoms to see the long-term clinical effects of the intervention.

ELIGIBILITY:
Inclusion Criteria for patient participants:

Clinical diagnosis of anxiety disorders (by psychiatrists using the structured clinical interview for DSM-IV-TR (SCID) with reference to the diagnostic criteria for GAD according to the ICD-10)

Exclusion Criteria for patient participants:

1. A history of serious cardiovascular, cerebrovascular diseases, stroke, or other neurological disorders, a history of gastrointestinal diseases.
2. Severe hearing or vision impairments.
3. Metallic implants in the body, such as non-removable dentures, stents, metal plates, joint metal replacements, etc.
4. Claustrophobia.
5. Acute or chronic diseases or infections.
6. Pregnancy or breastfeeding.
7. Smoking or drinking alcohol within 24 hours before the experiment.
8. Previous participation in similar experiments conducted by this institution.

Inclusion Criteria for healthy control participants:

1. No physical diseases or mental disorders.
2. No claustrophobia.
3. No hereditary diseases.
4. No medication history or smoking history.
5. Females not pregnant and not in their menstrual period.
6. Normal vision or corrected vision, no smoking, drinking alcohol, or taking medication within 24 hours prior to the experiment.
7. No previous participation in similar experiments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in participants' skin conductance response (SCR) | Baseline; every week (assessed weekly up to 8 weeks from the date of last intervention session)
  The level of SCR will be assessed for each experiment trial as the base-to-peak amplitude difference in skin conductance of the largest deflection (in micro-siemens; pS) in the 0.5-4.5-slatency window after stimulus onset.
Changes in the prefrontal cortex measured with fMRI | Baseline; once per week (assessed weekly up to 8 weeks from the date of last intervention session)
  Changes in the difference in blood oxygenation level dependent (BOLD) signals in the prefrontal cortex before and after the intervention.
Changes in the amygdala measured with fMRI | Baseline; once per week (assessed weekly up to 8 weeks from the date of last intervention session)
  Changes in the difference in blood oxygenation level dependent (BOLD) signals in the amygdala before and after the intervention.
Changes in the hippocampus measured with fMRI | Baseline; once per week (assessed weekly up to 8 weeks from the date of last intervention session)
  Changes in the difference in blood oxygenation level dependent (BOLD) signals in the hippocampus before and after the intervention.

SECONDARY OUTCOMES:
Changes in the State-Trait Anxiety Scale (STAI) | Baseline; once per week (assessed weekly up to 8 weeks from the date of last intervention session); 3 months (assessed at the week after 3 months from the last intervention session)
  The STAI assesses the current state of anxiety and relatively stable aspects of anxiety proneness, each subscale consisting of 20 items. Each item is rated on a 4-point Likert scale, ranging from "Not at all" to "Very much". Higher summed scores in subscales indicate greater state anxiety and trait anxiety.
Changes in the Intolerance of Uncertainty Scale-12 (IUS-12) | Baseline; once per week (assessed weekly up to 8 weeks from the date of last intervention session); 3 months (assessed at the week after 3 months from the last intervention session)
  The IUS measures individuals' emotional, cognitive, and behavioral responses or tolerance to uncertain situations, consisting 12 items. Each item is rated on a 5-point Likert scale, ranging from "Not at all characteristic of me" to "Entirely characteristic of me". Higher summed total scores suggest a higher level of intolerance of uncertainty.
Changes in the Anxiety Sensitivity Index (ASI) | Baseline; once per week (assessed weekly up to 8 weeks from the date of last intervention session); 3 months (assessed at the week after 3 months from the last intervention session)
  The ASI measures the extent to which individuals are sensitive to their own anxiety symptoms, consisting 12 items. Each item is rated on a 5-point Likert scale, ranging from "Not at all characteristic of me" to "Entirely characteristic of me". Higher summed total scores indicate greater anxiety sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Jingchu Hu, Dr., Principal Investigator — Shenzhen Kangning Hospital

IPD SHARING:
Plan to Share IPD: Yes
We will share our data on the Open Science Framework after data collection
Supporting Information: Study Protocol, SAP
Time Frame: The information will be shared after the related paper is published and will be available for at least one year.
Access Criteria: The information will be shared on the Open Science Framework for the public.